CLINICAL TRIAL: NCT00529581
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Titration Study to Assess the Safety, Tolerability, and Efficacy of C105 in Persons With Multiple Sclerosis With Cognitive Impairment
Brief Title: A Study of C105 on Cognitive Dysfunction in Persons With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cognition Pharmaceuticals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22029
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Cognition Disorders; Multiple Sclerosis
Keywords: multiple sclerosis; cognitive impairment; cognitive dysfunction; Cognitive Dysfunction associated with Multiple Sclerosis
MeSH Terms: conditions — Cognition Disorders; Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: C105

SUMMARY:
The purpose of this study is to determine the safety and efficacy of C105 in treating the cognitive deficits that can occur due to multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Males/females at least 18 years old and < 65 years old, capable of understanding and complying with the protocol, including speaking and writing fluent English and having at least a 9th grade education
* Clinically definite diagnosis per McDonald criteria of Multiple Sclerosis as confirmed by the Investigator (Relapsing-Remitting or Secondary Progressive)
* Stable disease and relapse-free for > 90 days as verified by Investigator
* Presence of cognitive deficit as measured score of -1.5 SD on the SDMT (oral version) or a score of -1.0 SD on the SDMT and -1.0 SD on either CVLT-II (total learning or delayed recall) or PASAT
* EDSS <= 6.5
* Standard score of >79 on the WRAT-4 Reading test
* Have given written informed consent prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care
* Capable of performing the requirements of a neuropsychological test battery including having at least 20/70 near visual acuity by near vision chart, with correction (i.e., eyeglasses) allowed
* If female, must neither be pregnant nor breast-feeding and she must either (a) be > 12 months post-menopausal or surgically sterilized or (b) must agree to use an acceptable method of birth control (including hormonal contraceptives, intra-uterine device, or barrier methods such as condoms, diaphragm, etc. with spermicide) for the duration of the study. Abstinence will not be considered an acceptable method of birth control.

Exclusion Criteria:

* Subjects with memory deficits caused by concomitant medication usage or other significant neurological/psychological disease, e.g., Alzheimer's disease, Parkinson's disease, stroke, TIA, Multi-infarct dementia, Huntington's disease, head trauma, or chronic CNS infection
* Evidence of other medical cause of dementia
* Evidence of Major Depressive Disorder as determined by a Beck Fast Screen core of >3 and clinician interview
* Use of the following medications: Antipsychotic agents, Centrally acting appetite suppression drugs (e.g., sibutramine), CNS stimulants or drugs that metabolize to them (e.g., amantadine, Concerta, methylphenidate, Adderall, ephedrine, selegiline), Strattera (atomoxetine), Tricyclic antidepressants (e.g., amitriptyline), Herbal preparations including Ginkgo Biloba or containing Ephedra or other stimulants, MAO inhibitors. Note: other medications may be excluded or permitted, depending on length of treatment and stability of dose
* Uncontrolled or labile hypertension, or any clinically significant, unstable, or major concomitant disorder as determined by the Principal Investigator
* Active malignancy within one year of study participation
* Known human immunodeficiency virus (HIV)
* Current diagnosis of unstable glaucoma
* History of myocardial infarction of symptomatic Coronary Artery Disease
* Evidence of ongoing ischemia or uncontrolled atrial or ventricular arrhythmias as shown by ECG
* History of epilepsy or other seizure disorders
* Clinically significant motor or speech residual neurological deficits (e.g., hemiparesis, aphasia) that interfere with completion of study procedures
* Baseline clinical laboratory values indicative of a clinically significant co-morbidity
* Significant recent history of (within past 12 months) or current drug or alcohol abuse (as defined by DSM-IV)
* Known allergy or hypersensitivity to amphetamines or other sympathomimetic amines
* Participation in any clinical trial with an investigational drug within 30 days prior to randomization
* In the opinion of the Principal Investigator should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test, Oral Version (SDMT) - Total # Correct | Change from baseline
Subject's Global Assessment of Cognitive Change | Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Munschauer, MD, Principal Investigator — SUNY Buffalo; Ralph Benedict, PhD, Principal Investigator — SUNY Buffalo
Locations (30):
- United States (30):
  - Saint Joseph's Hospital, Barrow Neurology Clinics, Phoenix, Arizona
  - Northwest Neuro Specialists, PLLC, Tuscon, Arizona
  - Research Center for Clinical Studies West, Lancaster, California
  - Loma Linda University, Department of Neurology, Loma Linda, California
  - Associated Neurologists, P.C., Danbury, Connecticut
  - Associated Neurologist of Southern Connecticut, PC, Fairfield, Connecticut
  - Yale University MS Center, New Haven, Connecticut
  - Neurology Associates, PA, Maitland, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Roskamp Institute, Sarasota, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Shepard Center, Atlanta, Georgia
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Health System, Department of Neurology, Detroit, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - The Jacobs Neurological Institute, Buffalo, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - MeritCare Neuroscience Clinic, Fargo, North Dakota
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Riverhills Healthcare, Inc, Cincinnati, Ohio
  - The Neurology Foundation, Inc., Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Integra Clinical Research, San Antonio, Texas
  - University of Virginia, Department of Neurology, Charlottesville, Virginia
  - Neurological Associates, Inc, Richmond, Virginia
  - Capitol Neurology, Charleston, West Virginia